CLINICAL TRIAL: NCT04942691
Title: Sport and Prevention of Bone Resorption
Brief Title: Prevention of Osteoporosis: Effects of Mini-trampoline Training on the Bone Remodeling
Acronym: TRAMBONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Patrizia Proia, Associate Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRAMP2021
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Perimenopausal Bone Loss; Postmenopausal Osteopenia
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The control group not performed physical activity during the time of the study. In the exercise group SuperJump® training was performed for three times a week, each session lasting 60 minutes for a total of 20-weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-exercise group (control group) (No Intervention): The control group not performed physical activity for a total of 20-weeks.
- exercise group (Experimental): The exercise group performed SuperJump® training that will be performed for three times a week, each session lasting 60 minutes for a total of 20-weeks.
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — training with trampoline. Each session lasted sixty minutes. Organization: a 5 minutes warm-up with breathing and mobility exercises from upper to lower body, central phase with jumping exercises involving the total body and 5 minutes of cool-down phase with total body active stretching exercise.
  Other Names: SuperJump® Training
  Arms: exercise group

SUMMARY:
The aim of the project is to study the effects on bone remodeling induced by training carried out with the trampoline in order to evaluate the reduction of the resorption itself and therefore the onset of osteoporosis in women.

DETAILED DESCRIPTION:
Bone mineral density is modified by various factors and in particular by diet, nutritional status and exercise recommended to preserve or increase bone mass in adults. The degree of bone formation and resorption can be assessed by measuring bone resorption markers in the blood or urine. To date, there is no information about the effect of training with an elastic trampoline on the reduction of bone resorption. The aim of the project is to study the effects on bone remodeling induced by training carried out with the trampoline, in order to evaluate the reduction of the resorption itself and therefore the onset of osteoporosis in women. To examine whether exercise affects bone remodeling, the C-terminal telopeptide bone resorption markers (CTX) and osteocalcin formation marker will be measured. For the evaluation of bone metabolism osteocalcin parathyroid hormone, Calcitonin, Vitamin D, Calcium, albumin, Phosphate, Potassium markers will be evaluated. The markers can be detected in serum. Women with no previous experience with the trampoline activity will participate in the project randomly assigned to the experimental training group (Jumpers) or to the control group, who will not do any training during the observation period (not Jumpers). The control group will be inserted in order to compare the data and further verify the efficiency of the treatment. Blood samples for bone resorption assay will be collected on the first day of training with the trampoline and 20 weeks. Each training session will be monitored by detecting heart rate (heart rate monitor) and subjective perception of fatigue (Borg scale). Each subject will be subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples thus obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Blood samples will be collected from the different groups of study. Samples will be analyzed and compared for Osteocalcin, parathyroid hormone, CTX, Calcitonin, Vitamin D Calcium, albumin, Phosphate, Potassium.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* age: 18-55 years
* currently injury free
* Body mass index between 18.5 and 28 kg/m2

Exclusion Criteria:

* bone fracture within the previous year
* use of medication or suffering from any condition known to affect bone metabolism
* pregnancy
* breastfeeding
* current smokers
* participation in moderate and high impact-activity for ≥3 h·week before enrolling the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Serum bone remodelling markers | 20 WEEKS
  bone resorption CTX and bone formation osteocalcin will be assessed at baseline and after 20weeks
Serum bone matabolism markers | 20 WEEKS
  PTH, calcitonin, Vitamin D, Calcium, Phosphate, Potassium will be assessed at baseline and after 20weeks
Plasma concentrations of Gastrointestinal peptides | 20 WEEKS
  GLP-1, GLP-2, GIP, PYY, Ghrelin will be assessed at baseline and after 20weeks

SECONDARY OUTCOMES:
body mass index (BMI) | 20 WEEKS
  Weight (Kg)
  Hight (m)
  BMI (kg/m2)
  All these measurements will be assessed at baseline and after 20weeks
body composition | 20 WEEKS
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 20weeks
insulin | 20 WEEKS
  measured in plasma will be assessed at baseline and after 20 weeks
glucose | 20 WEEKS
  measured in plasma will be assessed at baseline and after 20 weeks
triglicerises | 20 WEEKS
  measured in plasma will be assessed at baseline and after 20 weeks
HDL | 20 WEEKS
  measured in plasma will be assessed at baseline and after 20 weeks
Cholesterol | 20 WEEKS
  measured in plasma will be assessed at baseline and after 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Proia, PhD, Principal Investigator — Faculty of Sport and Physical Education, University of Palermo
Locations (1):
- Sport and Exercise Research Unit, Palermo University, Palermo, Italy

REFERENCES:
- [Derived] Vasto S, Amato A, Proia P, Caldarella R, Cortis C, Baldassano S. Dare to jump: The effect of the new high impact activity SuperJump on bone remodeling. A new tool to maintain fitness during COVID-19 home confinement. Biol Sport. 2022 Oct;39(4):1011-1019. doi: 10.5114/biolsport.2022.108993. Epub 2021 Dec 30. PMID 36247958